CLINICAL TRIAL: NCT06509048
Title: Effect of Combined Theta-gamma Frequency Subthalamic Nucleus Stimulation on Verbal Fluency in Parkinson Disease: a Randomized, Double-blind, Crossover Study
Brief Title: Combined Theta-gamma STN Stimulation for Verbal Fluency in Parkinson Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Maurizio Zibetti, Professor, University of Turin, Italy
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Theta-Gamma DBS
Record Dates: First submitted 2024-07-03; First posted 2024-07-19 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Parkinson Disease
Keywords: Deep brain stimulation; Verbal fluency; Parkinson's disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Stimulation (No Intervention): Standard STN-DBS stimulation
- Theta-Gamma Stimulation (Experimental): Standard STN-DBS stimulation with addiction of bilateral theta frequency stimulation of ventral contacts
  Interventions: Other: STN-DBS Theta Gamma Stimulation

INTERVENTIONS:
Other: STN-DBS Theta Gamma Stimulation — Standard STN-DBS stimulation with addiction of bilateral theta frequency stimulation of ventral contacts
  Arms: Theta-Gamma Stimulation

SUMMARY:
Deep Brain Stimulation (DBS) of the subthalamic nucleus (STN) is an established, effective, and relatively safe therapeutic option for Parkinson's disease (PD) patients presenting levodopa-related motor complications despite the best medical therapy . Chronic high-frequency (130-180 Hz) stimulation is known to reduce motor fluctuations and dyskinesia, and to improve quality of life and several non-motor symptoms . However, current evidence suggests a long term decline of cognitive performance in PD patients with STN-DBS compared to those without DBS, especially executive function processes including verbal fluency.

Preliminary evidence from pilot studies suggested that low frequency theta oscillations (4-10 Hz) within the STN and correlated cortical networks are important in cognition, including verbal fluency, color-word interference, and spatial and episodic memory; cortical structures involved in category verbal fluency encompass not only the prefrontal cortex, but also the hippocampus and related medial temporal structures. There is also evidence that theta STN stimulations lead to a worsening of motor symptoms, compared with no stimulation and therapeutic stimulation (gamma frequency).

To date, new DBS systems allow the use of multiple current sources and/or frequency settings at different depths and directions in a single electrode, and then to combine different stimulation frequencies.

Considering this, the aim is to evaluate the use of combined high (gamma) and very low (theta) frequency stimulation in a randomized, cross-over, double-blind trial with this principal research questions:

1. Can combined theta-gamma theta frequency STN stimulation improve verbal fluency in PD patients?
2. Can combined theta-gamma frequency STN stimulation improve verbal frequency without worsening cardinal motor symptoms?

DETAILED DESCRIPTION:
Each patient will receive two treatment periods, each lasting one month, in a randomized, cross-over, double-blind study design.

Patients will be randomly assigned to one of two sequences: Group 1 will receive standard DBS first followed by theta-gamma DBS, while Group 2 will receive theta-gamma DBS first followed by standard DBS. This design ensures that each patient serves as their own control, thereby reducing variability and enhancing the accuracy of the findings. A computer program will generate the randomization list.

One investigator, in charge of changing DBS parameter settings, will be unblinded to stimulation parameters and aware of the randomization sequence. The theta-gamma stimulation will be set maintaining the classical stimulation of the patient (gamma frequency, 100-180 Hz), with bilateral addiction of a ventral contact for stimulation with theta frequency (4-10 Hz).

Two investigators, blinded to stimulation parameters and randomization sequence, will conduct clinical and neuropsychological assessments.

The unblinded investigator will decide on a possible switch to the next sequence if the symptoms will not be well tolerated by the patient. In case of persistent worsening even after the second modification, the patient will be dropped out from the study. Dopaminergic therapy will be stable during the study course.

The clinical and neuropsychological test battery will include: motor state, evaluated with the Movement Disorder Society - Unified Parkinson Disease Rating Scale (MDS-UPDRS); Cognitive screening test, as per Mini Mental State Examination (MMSE); Beck Depression Inventory - Short Form (BDI-SF); Questionnaire for Impulsive-Compulsive Disorders in Parkinson's Disease-Rating Scale (QUIP-RS); Phonemic and semantic verbal fluency test (letter, episodic category, non-episodic category, and category switching).

The neuropsychological test battery will be conducted at baseline and at the end of first and second month of evaluation. The verbal fluency evaluation will be conducted also one hour after the change of stimulation parameters, to also evaluate its impact at a short time distance.

The evaluation will be conducted in the morning, during the ON phase, in order to avoid possible effects of wearing-off on cognitive performance.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old,
* Optimized DBS therapy in the last month,
* Stable medication regimen in the last month
* Able to provide informed consent
* Fluent in Italian
* Able to complete cognitive testing
* Patients implanted with bilateral Vercise Cartesia™ Directional Leads in the STN connected to a Vercise™ or Vercise Gevia™ or Vercise Genus™ DBS system

Exclusion Criteria:

* History of dementia (MMSE ≤ 25),
* Major substance abuse,
* Stimulation provided in the more ventral contact

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-11-10 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Verbal Fluency - Phonemic Fluency | Baseline; 1st month; 2nd month
  Number of words per three given letters in one minute for each letter
Verbal Fluency - Semantic Fluency - Episodic category | Baseline; 1st month; 2nd month
  Number of words per episodic category (related to personal past experiences, e.g., "memorable events" or "significant places") in one minute
Verbal Fluency - Semantic Fluency - Non-episodic category | Baseline; 1st month; 2nd month
  Number of words per non episodic category (belonging to a specific category, e.g., animals, fruits) in one minute
Verbal Fluency - Semantic Fluency - Switching | Baseline; 1st month; 2nd month
  Number of words with switch of categories: participants are required to alternately generate words from two different non episodic categories (e.g., animals and fruits) in one minute
Motor symptoms | Baseline; 1st month; 2nd month
  Movement Disorder Society - Unified Parkinson Disease Rating Scale part III (MDS-UPDRS III). Change in total MDS UPDRS part III score between standard and Theta-Gamma stimulation. Score range: 0-132 (higher score indicates worse motor performance)

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Zibetti, Principal Investigator — AOU Città della Salute e della Scienza Torino
Locations (1):
- AOU Città della Salute e della Scienza Torino, Torino, Italy

IPD SHARING:
Plan to Share IPD: No